CLINICAL TRIAL: NCT06791031
Title: PCSK9 inhibitoRs for Early Passivation of coRonary athEroSclerotic plaqueS in Acute Coronary Syndromes (REPRESS): Study Protocol for a Multicenter Randomized Controlled Trial
Brief Title: PCSK9 inhibitoRs for Early Passivation of coRonary athEroSclerotic plaqueS in Acute Coronary Syndromes (REPRESS)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Yong He, Professor, Sichuan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WestChinaH-CVD-009
Record Dates: First submitted 2025-01-11; First posted 2025-01-24 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2024-11

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "PCSK9i early" intensified therapy group (Experimental): Initial addition of PCSK9i to moderate-intensity statin
  Interventions: Drug: PCSK9 inhibitor (PCSK9i)
- Guideline-directed medical therapy group (No Intervention): Stepwise lipid-lowering strategies based on the 2025 American College of Cardiology/American Heart Association guidelines for ACS, Chinese Lipid Management Guidelines (2023), and Expert Consensus on Clinical Pathways for Lipid Management in Chinese Patients with ACS.

INTERVENTIONS:
Drug: PCSK9 inhibitor (PCSK9i) — Patients randomized to the "PCSK9i early" intensified therapy group will receive initial treatment with a PCSK9 inhibitor-either evolocumab 140 mg or alirocumab 75 mg, both administered subcutaneously every two weeks with the initial dose given during hospitalization and subsequent doses self-administered at home-or inclisiran sodium 300 mg (equivalent to 284 mg inclisiran), administered by healthcare professionals at baseline and again at the 3-month study visit. All patients will receive moderate-intensity statin, including atorvastatin 20 mg or rosuvastatin 10 mg. The intervention will be initiated during hospitalization for the index ACS event, within 24 hours of randomization, irrespective of baseline LDL-C levels or prior statin use.
  Arms: "PCSK9i early" intensified therapy group

SUMMARY:
In this prospective, multicenter, open-label trial, 212 ACS patients will be randomized 1:1 to either the "PCSK9i early" intensified therapy group (initial addition of PCSK9i to moderate-intensity statin) or the guideline-directed medical therapy group for 6 months. Serial OCT imaging of non-culprit arteries (20-70% stenosis) is performed at baseline and 6 months. The primary endpoint is the absolute change in minimum fibrous cap thickness at 6 months, and secondary endpoints including changes in lumen area, lipid arc, macrophage infiltration, LDL-C reduction, and target LDL-C achievement.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age ≥ 18 years at screening
* Acute coronary syndrome who underwent PCI of the culprit lesions.
* Non-culprit vessel (target vessel) meets the following criteria after culprit vessel PCI:
* Target vessel diameter > 2.5 mm, suitable for OCT examination
* Target vessel with angiographically estimated stenosis (diameter stenosis 20-70%)
* Target vessel must be native coronary arteries, vessel segment without previous PCI
* Target vessel cannot be a venous or arterial bridge vessel
* Ability to cooperate the requirements of the study and to offer written informed consent
* Willingness to complete follow-up visits and examinations as required by the schedule
* Life expectancy > 1 year

Exclusion Criteria:

* Left main disease of non-culprit artery, defined as ≥ 50% reduction in lumen diameter of the left main coronary artery via angiographic visual estimation
* Thrombotic target lesion, severe calcification or tortuosity lesions unfavorable for OCT examination
* Coronary artery anatomy that prevents complete imaging of the segment of interest (including at least 5 mm of both edges of the stenosis)
* True bifurcation lesions requiring stenting
* TIMI flow < 2 of the culprit-related arteries after PCI
* Unstable clinical status (cardiogenic shock, hemodynamic or electrical instability)
* Advanced heart failure (New York cardiac class III-IV)
* Ischaemic stroke within the past 6 months or cerebral haemorrhage at any time in the past
* Severe valvular disease or valvular disease that may require surgery or percutaneous valve replacement
* Diffuse coronary artery lesions or the presence of ≥ 1 untreated non-culprit lesion (non-culprit flow-restricting lesion planned for near-term, phase II PCI)
* Target vessel with coronary artery bypass grafting or PCI
* Planned major surgery requiring interruption of dual-antiplatelet therapy
* Statin intolerance and patients unsuitable for statin therapy with alanine aminotransferase greater than 3 times the upper limit of normal or creatine kinase greater than 3 times the upper limit of normal (not attribute to an acute MI) or greater
* Familial hypercholesterolaemia
* Prior (within 180 days prior to the first study visit) exposure to PCSK9i, either as an experimental or marketed drug
* Female subjects of childbearing potential, defined as all female subjects who are physiologically capable of becoming pregnant, unless such female subjects are using an effective method of contraception during the trial
* Women who are pregnant or breastfeeding or intend to become pregnant
* Comorbidities with malignancies, active infections, or major hematologic, metabolic, or endocrine disorders are judged unsuitable by the investigator
* Severe hepatic insufficiency (Child-Pugh class C)
* Severe renal dysfunction (estimated glomerular filtration rate < 30 mL/min/1.73 m2)
* Current enrollment in another investigational device or drug study
* Poor adherence and unable to complete the expected follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Absolute change in the minimum fibrous cap thickness of target lesions | At 6 months post randomization
  Absolute change in the minimum fibrous cap thickness of target lesions from baseline to 6 months.

SECONDARY OUTCOMES:
Percent change in minimum fibrous cap thickness of target vessels | At 6 months post randomization
  Percent change in minimum fibrous cap thickness of target vessels from baseline to 6 months.
Absolute change in mean minimum fibrous cap thickness across target vessels | At 6 months post randomization
  Absolute change in mean minimum fibrous cap thickness across target vessels from baseline to 6 months.
Absolute changes in minimum lumen area of target vessels | At 6 months post randomization
  Absolute changes in minimum lumen area of target vessels from baseline to 6 months.
Absolute changes in maximum lipid arc of target vessels | At 6 months post randomization
  Absolute changes in maximum lipid arc of target vessels from baseline to 6 months.
Presence of macrophage infiltration in target vessels | At 6 months post randomization
  Presence of macrophage infiltration in target vessels from baseline to 6 months.
Proportion of patients with OCT-identified vulnerable plaques | At 6 months post randomization
  Proportion of patients with OCT-identified vulnerable plaques (defined as FCT < 75 µm plus at least two of three features: lipid arc > 180°, MLA < 3.5 mm², and macrophage infiltration) from baseline to 6 months.
Change in total cholesterol | At 3 months and 6 months post randomization
  Change in total cholesterol from baseline to 3 and 6 months.
Change in apolipoprotein B | At 3 months and 6 months post randomization
  Change in apolipoprotein B from baseline to 3 and 6 months.
Change in lipoprotein(a) | At 3 months and 6 months post randomization
  Change in lipoprotein(a) from baseline to 3 and 6 months.
Change in triglycerides | At 3 months and 6 months post randomization
  Change in triglycerides from baseline to 3 and 6 months.
Change in very low-density lipoprotein cholesterol | At 3 months and 6 months post randomization
  Change in very low-density lipoprotein cholesterol from baseline to 3 and 6 months.
Change in low-density lipoprotein cholesterol | At 3 months and 6 months post randomization
  Change in low-density lipoprotein cholesterol from baseline to 3 and 6 months.
Change in high-density lipoprotein cholesterol | At 3 months and 6 months post randomization
  Change in high-density lipoprotein cholesterol from baseline to 3 and 6 months.
Proportion of patients achieving predefined LDL-C targets | At 3 months and 6 months post randomization
  Proportion of patients achieving predefined LDL-C targets (< 1.4 mmol/L) from baseline to 3 and 6 months.
Adherence to lipid-lowering therapy | At 3 months and 6 months post randomization
  Adherence (proportion of days covered) to lipid-lowering therapy (statin, cholesterol absorption inhibitor, and PCSK9i) from baseline to 3 months and 6 months.

OTHER OUTCOMES:
Incidence of major adverse cardiovascular events (MACEs) | At 6 months and 12 months post randomization
  MACEs are defined as the composite of cardiac death, nonfatal myocardial infarction, nonfatal stroke, and ischemia-driven revascularization.
Incidence of bleeding events | At 6 months and 12 months post randomization
  Bleeding events are defined according to the Academic Research Consortium (ARC) criteria.
Change in high-sensitivity C-reactive protein | At 3 months and 6 months post randomization
  Change in high-sensitivity C-reactive protein from baseline to 3 and 6 months.
Change in Interleukin-6 (IL-6) | At 3 months and 6 months post randomization
  Change in IL-6 levels from baseline to 3 and 6 months.
Change in tumor necrosis factor-alpha (TNF-α) | At 3 months and 6 months post randomization
  Change in TNF-α levels from baseline to 3 and 6 months.
Change in absolute T-cell count | At 3 months and 6 months post randomization
  Change in absolute T-cell count from baseline to 3 and 6 months.
Change in absolute B-cell count | At 3 months and 6 months post randomization
  Change in absolute B-cell count from baseline to 3 and 6 months.
Change in absolute natural killer (NK) cell count | At 3 months and 6 months post randomization
  Change in absolute NK cell count from baseline to 3 and 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Yong He, Principal Investigator — Department of Cardiology, West China Hospital of Sichuan University

IPD SHARING:
Plan to Share IPD: Yes
IPD that will be shared include anonymized data on baseline characteristics, primary and secondary outcome measures.